CLINICAL TRIAL: NCT00457418
Title: A Pharmacokinetic Study of PEG-Intron, Administered Weekly in Subjects With High-Risk Melanoma
Brief Title: High-Dose PEG-Intron Pharmacokinetic Study in Patients With Melanoma (Study P04831 AM2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04831
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — peginterferon alfa-2b

ARMS (1):
- PEG-Intron (Experimental): 6 ug/kg/week, SC (first 8 weeks)
  3 ug/kg/week, SC (252 weeks [weeks 9-260], maintenance)
  Interventions: Drug: PEG-Intron

INTERVENTIONS:
Drug: PEG-Intron
  Other Names: SCH 054031; peginterferon alfa-2b

SUMMARY:
The purpose of this study is to establish the pharmacokinetics of PEG-Intron, administered at a dose of 6 μg/kg/week for 8 weeks (induction treatment), followed by a dose of 3 μg/kg/week for up to 252 weeks (maintenance treatment), in patients with high risk melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years of age, of either sex, and of any race.
* Cytologically or histologically-confirmed melanoma, arising from a cutaneous or unknown site of origin, at Stages IIB, IIC, IIIA, IIIB, IIIC according to the American Joint Committee on Cancer (AJCC) 2001 guidelines.
* Adequate hepatic, renal and bone marrow function within 4 weeks prior to initiation of study treatment.
* Subjects presenting with synchronous primary and regional melanoma must have had adequate surgical margins surrounding the primary lesion.
* Full lymphadenectomy must be performed within 90 days prior to initiation of study treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Give informed consent according to International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) and national/local policy.
* Be able to adhere to dose and visit schedules.
* Female subjects of childbearing potential must be using a medically accepted method of birth control prior to Screening and agree to continue its use during the study or be surgically sterilized.
* Female subjects of childbearing potential must have a negative serum pregnancy test at Screening.

Exclusion Criteria:

* Female subjects who are pregnant, intend to become pregnant, or are breastfeeding.
* Previous treatment with interferon alpha, chemotherapy or immunotherapy for melanoma.
* Ocular melanoma, or melanoma of the mucous membranes.
* Evidence of distant or non-regional lymph node metastases.
* In-transit melanoma, even if the lesion has been resected.
* Disease that cannot be completely surgically resected.
* Lack of recovery from recent surgery.
* Prior malignancy within the past 5 years, except surgically cured squamous cell carcinoma of the skin, successfully resected early stage cutaneous melanoma, or cervical carcinoma in situ.
* Severe cardiovascular disease.
* Thyroid dysfunction not responsive to therapy.
* Uncontrolled diabetes mellitus (in the opinion of the investigator).
* Active autoimmune disease.
* Active and/or uncontrolled infection.
* History of seropositivity for human immunodeficiency virus (HIV).
* Pre-existing psychiatric condition.
* Clinical diagnosis of substance abuse of one or more of the following drugs within the following timeframes (excluding time spent in detoxification, hospitalization or incarceration):

  * Alcohol, intravenous drug use, inhalational, psychotropics, narcotics, cocaine, prescription or over-the-counter drugs: within 1 year of the Screening visit.
  * Methadone, buprenorphine hydrochloride (HCl), and/or butorphanol tartrate: within 1 year of Screening visit, unless subject has drug screen negative for other (non-narcotic) drugs documented in the past year and repeated negative within 2 months of Screening visit.
  * Multi-drug abuse (2 or more substances in 16a and 16b): within 3 years of Screening visit.
  * Marijuana:

    * If historic use is deemed excessive by the principal investigator (or medically qualified individual), or is interfering with the subject's life, then the subject is not eligible and should not be screened.
    * If marijuana use is not deemed excessive by principal investigator and does not interfere with life, subject must discontinue any current use of marijuana prior to entry into study.
* Medical condition requiring chronic systemic corticosteroids.
* Known allergy to the drug substance or any of the excipients in the PEG-Intron formulation.
* Any situation or condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Use of any investigational drugs within 30 days of study entry.
* Participation in other clinical studies of investigational treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-02-20 (Actual); Primary Completion 2008-05-27 (Actual); Study Completion 2012-07-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Daud AI, Xu C, Hwu WJ, Urbas P, Andrews S, Papadopoulos NE, Floren LC, Yver A, Deconti RC, Sondak VK. Pharmacokinetic/pharmacodynamic analysis of adjuvant pegylated interferon alpha-2b in patients with resected high-risk melanoma. Cancer Chemother Pharmacol. 2011 Mar;67(3):657-66. doi: 10.1007/s00280-010-1326-9. Epub 2010 May 28. PMID 20509027

RESULTS

PARTICIPANT FLOW:
Period: Pharmacokinetic (PK) Sampling Phase
Arm/Group | PEG-Intron
Started | 32
Completed | 27
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Progression of Disease | 1
Not completed — Non-compliance with protocol | 2
Period: Post PK Maintenance
Arm/Group | PEG-Intron
Started | 31 (4 participants didn't complete the PK sampling phase but continued to post PK maintenance treatment.)
Completed | 3
Not Completed | 28
Not completed — Adverse Event | 10
Not completed — Progression of Disease | 6
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | PEG-Intron
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of PEG-Intron at 12 Weeks
Description: AUC was defined as the actual body exposure to drug after administration of a dose of the drug.
Time Frame: Predose, and 24, 48, 72, 96, and 168 hours postdose at 12 weeks
Population: Participants who completed the full 12 weeks of treatment without any significant dose modification (dose reduction or missing dose)
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | PEG-Intron
Number analyzed (Participants) | 20
pg*hr/mL | 235000 (56400) [207592 to 251430]

2. Primary Outcome: Maximum Serum Concentration (Cmax) of PEG-Intron at 12 Weeks
Description: Cmax was defined as observed maximum plasma concentration.
Time Frame: Predose, and 24, 48, 72, 96, and 168 hours postdose at 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PEG-Intron
Number analyzed (Participants) | 20
pg/mL | 2620 (865) [2173 to 2829]

3. Primary Outcome: Average Concentration Within the Dosing Interval (Cavg) of PEG-Intron at 12 Weeks
Description: Cavg was defined as average plasma concentration.
Time Frame: Predose, and 24, 48, 72, 96, and 168 hours postdose at 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PEG-Intron
Number analyzed (Participants) | 20
pg/mL | 1400 (336) [1236 to 1497]

4. Primary Outcome: Minimum Serum Concentration (Cmin) of PEG-Intron at 12 Weeks
Description: Cmin was defined as observed minimum plasma concentration.
Time Frame: Predose, and 24, 48, 72, 96, and 168 hours postdose at 12 weeks
Population: There were 19 evaluable participants (20 participants completed the full 12 weeks of treatment without any significant dose modification and there was no concentration data for 1 participant at Week 12).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PEG-Intron
Number analyzed (Participants) | 19
pg/mL | 626 (269) [498 to 678]

5. Primary Outcome: Observed Time to Achieve Cmax (Tmax) of PEG-Intron at 12 Weeks
Description: Tmax was defined as time of maximum plasma concentration.
Time Frame: Predose, and 24, 48, 72, 96, and 168 hours postdose at 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | PEG-Intron
Number analyzed (Participants) | 20
hours | 24.00 [24.00 to 48.00]

6. Primary Outcome: Apparent Clearance(CL/F) of PEG-Intron at 12 Weeks
Description: CL/F was defined apparent clearance - the volume of plasma in the vascular compartment cleared of drug per unit of time and per kilogram of body weight by the processes of metabolism and excretion.
Time Frame: Predose, and 24, 48, 72, 96, and 168 hours postdose at 12 weeks
Population: There were 15 evaluable participants (20 participants completed the full 12 weeks of treatment without any significant dose modification but for 5 participants CL/F could not be reported because t1/2 could not be accurately determined).
Measure: Mean (Standard Deviation); unit: L/hr/kg
Arm/Group | PEG-Intron
Number analyzed (Participants) | 15
L/hr/kg | 0.0129 (0.00284)

7. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) was defined as any untoward medical occurrence or unfavorable and unintended sign in a subject administered a pharmaceutical product, biologic (at any dose), or medical device, whether or not considered related to the use of that product.
Time Frame: Entire study duration (up to 5 years)
Measure: Number; unit: participants
Arm/Group | PEG-Intron
Number analyzed (Participants) | 32
participants | 32

ADVERSE EVENTS:
Arm/Group | PEG-Intron
Serious Adverse Events (participants affected / at risk) | 9/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron (N=32)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
GLAUCOMA (Eye disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1)
APPENDICITIS PERFORATED (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron (N=32)
ANAEMIA (Blood and lymphatic system disorders) | 2 (3)
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (14)
NEUTROPENIA (Blood and lymphatic system disorders) | 7 (31)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
EAR PAIN (Ear and labyrinth disorders) | 2 (3)
HYPOTHYROIDISM (Endocrine disorders) | 3 (3)
DRY EYE (Eye disorders) | 3 (3)
VISION BLURRED (Eye disorders) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (7)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 4 (5)
DIARRHOEA (Gastrointestinal disorders) | 20 (33)
DRY MOUTH (Gastrointestinal disorders) | 3 (3)
FLATULENCE (Gastrointestinal disorders) | 2 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 23 (41)
VOMITING (Gastrointestinal disorders) | 8 (13)
CHEST PAIN (General disorders) | 2 (2)
CHILLS (General disorders) | 26 (39)
FATIGUE (General disorders) | 29 (52)
INFLUENZA LIKE ILLNESS (General disorders) | 6 (8)
INJECTION SITE RASH (General disorders) | 2 (2)
INJECTION SITE REACTION (General disorders) | 13 (15)
MUCOSAL INFLAMMATION (General disorders) | 2 (3)
OEDEMA (General disorders) | 4 (4)
PAIN (General disorders) | 2 (2)
PYREXIA (General disorders) | 27 (44)
BRONCHITIS (Infections and infestations) | 2 (2)
LOCALISED INFECTION (Infections and infestations) | 2 (2)
SINUSITIS (Infections and infestations) | 3 (6)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 (11)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 (5)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 2 (5)
NEUTROPHIL COUNT DECREASED (Investigations) | 11 (25)
PLATELET COUNT DECREASED (Investigations) | 3 (5)
WEIGHT DECREASED (Investigations) | 3 (3)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 8 (26)
DECREASED APPETITE (Metabolism and nutrition disorders) | 27 (33)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (4)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 13 (43)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (8)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (9)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 18 (24)
DIZZINESS (Nervous system disorders) | 5 (5)
DYSGEUSIA (Nervous system disorders) | 3 (3)
HEADACHE (Nervous system disorders) | 23 (48)
SOMNOLENCE (Nervous system disorders) | 5 (6)
AGITATION (Psychiatric disorders) | 2 (3)
ANXIETY (Psychiatric disorders) | 7 (7)
DEPRESSION (Psychiatric disorders) | 12 (12)
INSOMNIA (Psychiatric disorders) | 9 (11)
MENTAL STATUS CHANGES (Psychiatric disorders) | 2 (2)
MOOD ALTERED (Psychiatric disorders) | 4 (5)
DYSURIA (Renal and urinary disorders) | 2 (2)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 5 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (15)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (6)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 (2)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 4 (4)
PRURITUS (Skin and subcutaneous tissue disorders) | 7 (7)
RASH (Skin and subcutaneous tissue disorders) | 10 (20)
HYPERTENSION (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator (PI) agrees not to publish/present any interim results of the study without Sponsor's prior written consent. The PI further agrees to provide to the sponsor 30 days prior to submission, review copies. The sponsor shall have editorial rights and the right to review and comment. If the parties disagree, PI agrees to meet with the sponsor's representatives for the purpose of making good faith efforts to discuss and resolve any such issues or disagreement.